CLINICAL TRIAL: NCT07083232
Title: Comparative Study on the Effect of Sitagliptin, Pioglitazone and Dapagliflozine on Myocardial Infarction Induced Experimentally in Diabetic Rats
Brief Title: The Effect of Sitagliptin, Pioglitazone and Dapagliflozine on Myocardial Infarction in Diabetic Rats
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, El Shazly Abdelaal Mohaseb, Assistant lecturer of pharmacology, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MD/AZ.AST./PHA006/8/231/5/2024
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2023-07

CONDITIONS: Diabetic; Myocardial Infarction
Keywords: Myocardial Infarction; Diabetic; Rats; Sitagliptin; Pioglitazone; Dapagliflozine
MeSH Terms: conditions — Myocardial Infarction | interventions — Streptozocin; Sitagliptin Phosphate; lactitol; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- standard normal diet and water group (Placebo Comparator): Group I: formed of normal animals. They were allowed standard normal diet and water. They received no drugs.
  Interventions: Dietary Supplement: standard normal diet
- low dose Streptozotocin group (Experimental): Group II: Non-treated diabetic rats; diabetes was induced by administration of 20% fructose solution in drinking water for 2 weeks, then intra peritoneal injection of a low dose STZ (40 mg/kg b.w.)
  Interventions: Drug: low dose Streptozotocin
- Sitagliptin group (Experimental): Group III: Sitagliptin treated diabetic group sitagliptin was administered by gastric gavage in a dose 10mg/ kg /day for 4 weeks
  Interventions: Drug: Sitagliptin (Novartis, USA)
- Pioglitazone group (Experimental): Group IV : Pioglitazone treated diabetic group ; Pioglitazone was administered by gastric gavage in a dose 10 mg/ kg /day for 4 weeks
  Interventions: Drug: Pioglitazone hydrochloride (Unipharma., Egypt)
- Dapagliflozine group (Experimental): Group V : Dapagliflozine treated diabetic group (G5); Dapagliflozine was administered by gastric gavage in a dose 1mg/ kg /day for 4 weeks
  Interventions: Drug: Dapagliflozine hemihydrate (Janssen, USA)

INTERVENTIONS:
Dietary Supplement: standard normal diet — Group I: formed of normal animals. They were allowed standard normal diet and water. They received no drugs
  Arms: standard normal diet and water group
Drug: low dose Streptozotocin — Non-treated diabetic rats; diabetes was induced by administration of 20% fructose solution in drinking water for 2 weeks, then intra peritoneal injection of a low dose STZ (40 mg/kg b.w.), was done
  Arms: low dose Streptozotocin group
Drug: Sitagliptin (Novartis, USA) — Sitagliptin treated diabetic group sitagliptin was administered by gastric gavage in a dose 10mg/ kg /day for 4 weeks
  Arms: Sitagliptin group
Drug: Pioglitazone hydrochloride (Unipharma., Egypt) — Pioglitazone treated diabetic group (G4); Pioglitazone was administered by gastric gavage in a dose 10 mg/ kg /day for 4 weeks
  Arms: Pioglitazone group
Drug: Dapagliflozine hemihydrate (Janssen, USA) — Dapagliflozine treated diabetic group (G5); Dapagliflozine was administered by gastric gavage in a dose 1mg/ kg /day for 4 weeks
  Arms: Dapagliflozine group

SUMMARY:
The aim of the present study is to evaluate the prophylactic effect of Sitagliptin, Pioglitazone and Dapagliflozine on Isoprenaline induced myocardial infarction in type II diabetic rats.

DETAILED DESCRIPTION:
The American Diabetes Association defined diabetes mellitus as a group of metabolic diseases characterized by hyperglycemia resulting from defects in insulin secretion, insulin action or both. The chronic hyperglycemia of diabetes is associated with long-term damage, dysfunction and failure of different organs, especially the eyes, kidneys, nerves, heart and blood vessels.

Myocardial ischemia represents a condition of sufferance for cardiomyocytes due to coronary blood flow reduction as compared to their metabolic needs, and it may exhibit through several clinical conditions.

People with type 2 diabetes mellitus are at increased risk of cardiovascular disease, heart failure and death, as compared with the general population. Studies show that the excess risks associated with diabetes mellitus are mediated primarily by hyperglycemia and overall poor risk factor control. Effective treatment of traditional cardiovascular risk factors has reduced the excess risk of atherosclerotic cardiovascular disease , such as acute myocardial infarction and stroke in people with type 2 diabetes mellitus.

In the last two decades, several studies have demonstrated reductions in the risk of cardiovascular outcomes and mortality in patients with type 2 diabetes mellitus with improved glucose and cholesterol-lowering therapies. Nevertheless, macrovascular disease remains the most common cause of death in type 2 diabetes mellitus patients and new diabetes therapies are highly desired, especially if they can offer cardiovascular benefits.

Sitagliptin is a potent and highly selective dipeptidyl peptidase-4 competitive inhibitor that does not affect the closely related enzymes dipeptidyl peptidase-8 or dipeptidyl peptidase-9 at therapeutic concentrations.

Sitagliptin found to enhance circulating glucagon-like peptide-1 levels through inhibition of dipeptidyl peptidase -IV activity.

which, in turn, provides cardiovascular protection probably through the anti-inflammatory and anti-atherosclerotic activities of glucagon-like peptide-1. Reduces blood glucose levels, in either the postprandial or the fasting state.

Multiple studies have suggested that pioglitazone, a peroxisome proliferatoractivated receptor γ agonist, used as an insulin-sensitizing agent in the treatment of type 2 diabetes mellitus , may have anti-atherosclerotic effects.

The mechanism of action of dapagliflozine influences a number of cardiovascular disease risk factors, in particular, decreasing blood pressure, reducing body weight (predominantly through reductions in total body fat mass, including visceral adipose tissue), reducing waist circumference, and lowering albuminuria and serum uric acid levels, with allow intrinsic risk of hypoglycemia.

Isoprenaline is a potent β-adrenergic agonist, increases the myocardial oxygen demand by mixture of its positive inotropic and chronotropic actions. Administration of isoprenaline in high doses to animals produces infarct like lesions in the heart similar to those present in myocardial infatction in humans.

The aim of the present study is to evaluate the prophylactic effect of Sitagliptin, Pioglitazone and Dapagliflozine on Isoprenaline induced myocardial infarction in type II diabetic rats.

ELIGIBILITY:
Inclusion Criteria:

* 50 adult male albino rats obtained from (Experimental Animal Breeding Farm, assuit -Cairo) weighing between 150- 200 g (at the beginning of the study)

Exclusion Criteria:

* Female rats --Weight >200g

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
blood glucose | one week

SECONDARY OUTCOMES:
tumor necrosis factor-α | One week

CONTACTS AND LOCATIONS:
Locations (1):
- Alazher University.assuit Branch, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol